CLINICAL TRIAL: NCT04160637
Title: Early Postoperative Serum Parathyroid Hormone Levels as a Predictor of Hypocalcaemia After Total Thyroidectomy: A Prospective Non-Randomized Study
Brief Title: Is There Benefit From Early Postoperative PTH Monitoring?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Sestre Milosrdnice (Other)
Responsible Party: Principal Investigator, Andro Košec, MD, PhD, Consultant Otorhinolaryngologist and Head and Neck Surgeon, University Hospital Sestre Milosrdnice
Other Study IDs: EP-PTH01
Record Dates: First submitted 2019-11-09; First posted 2019-11-13 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Hypocalcemia; Thyroid; Postoperative Complications; Parathyroid Dysfunction; Hormone Disturbance
Keywords: parathyroid hormone; total thyroidectomy; hypocalcemia; postoperative; predictive factor
MeSH Terms: conditions — Hypocalcemia; Thyroid Diseases; Postoperative Complications; Parathyroid Diseases; Endocrine System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with post-thyroidectomy hypocalcemia: Patients with postoperative hypocalcemia defined as serum calcium levels < 2.00 mmol/L regardless of clinical symptoms present. Patients may have low or normal PTH range (defined by the Department of Laboratory Diagnostics reference range from 1.6 to 6.9 pmol/L)
  Interventions: Diagnostic Test: Immediate postoperative PTH serum sampling and cut-off value identification
- Patients without post-thyroidectomy hypocalcemia: Patients without postoperative hypocalcemia defined as serum calcium levels > 2.00 mmol/L regardless of clinical symptoms present. Patients may have low or normal PTH range (defined by the Department of Laboratory Diagnostics reference range from 1.6 to 6.9 pmol/L)
  Interventions: Diagnostic Test: Immediate postoperative PTH serum sampling and cut-off value identification

INTERVENTIONS:
Diagnostic Test: Immediate postoperative PTH serum sampling and cut-off value identification — The patients will undergo immediate post-thyroidectomy PTH sampling in order to establish a cut-off value for identifying patients at risk for postoperative hypocalcemia within the first 5 postoperative days.

SUMMARY:
This study is designed as a prospective non-randomized longitudinal single-center cohort study. It will enroll around 120 patients undergoing total thyroidectomy with data being collected from September 2019 up to December 2019. The hypothesis is that a significant association and cut-off point in PTH levels may be established with regard to postoperativne hypocalcaemia.

Primary outcome measures are presence of hypocalcemia on the first and fifth postoperative day. Secondary outcome measures are the need for calcium supplement therapy during the first five postoperative days and amount of medication given.

Associations between variables will be assessed using Spearman's rho rank correlation coefficient, the Kruskal-Wallis test for independent samples and a logistic regression model to test statistically significant correlations between PTH and serum calcium values as a primary end point.

DETAILED DESCRIPTION:
This study is designed as a prospective non-randomized longitudinal single-center cohort study. It will enroll around 120 patients undergoing total thyroidectomy with data being collected from September 2019 up to December 2019. The study was approved by the Hospital Board of Ethics, according to the Declaration of Helsinki Ethical Principles for Medical Research Involving Human Subjects, adopted by the 18th World Medical Assembly, Helsinki, Finland, June 1964, and as amended most recently by the 64th World Medical Assembly, Fontaleza, Brazil, October 2013. The patients will be eligible if they undergo total thyroidectomy regardless of the surgical indication, if complete serum PTH and calcium data are available through the first five postoperative days and if they sign an informed consent form. Patients with incomplete data, preoperative pathological calcium or PTH levels, or suffering from conditions affecting calcium metabolism and parathyroid function will be excluded from the study.

Demographic and clinical data including age, sex, preoperative and postoperative laboratory values (serum calcium and PTH), neck dissection procedures, and postoperative calcium supplement therapy will be noted. Primary outcome measures are presence of hypocalcemia on the first and fifth postoperative day. Secondary outcome measures are the need for calcium supplement therapy during the first five postoperative days and amount of medication given. Preoperative blood samples for serum PTH and calcium measurements will be obtained after hospital admission. Postoperative serum PTH will be sampled 1 hour after surgery and at 7 am on the first and fifth postoperative day. Serum calcium sampling will be performed daily if a patient has hypocalcemia detected on the first postoperative day. Hypocalcemia is defined as serum calcium levels < 2.00 mmol/L regardless of clinical symptoms present. Normal PTH range is defined by the Department of Laboratory Diagnostics reference range - from 1.6 to 6.9 pmol/L. The recovery of parathyroid function is defined as the return of serum PTH and serum calcium to normal values, requiring no further calcium or vitamin D supplementation. If the patient does not have laboratory or clinical signs of hypocalcemia, calcium supplement therapy will not be administered. Supplement therapy will be administered in patients with laboratory findings confirming hypocalcemia. Supplement therapy consists of either peroral elemental calcium (calcium carbonate, 1-gram unit) or calcitriol (0.5 microgram unit) or both. If postoperative calcium and PTH are normal and there are no symptoms of discomfort, the patient will be discharged on the first or second postoperative day and serum PTH and calcium sampling will be performed on an outpatient basis. If the patient did not receive treatment during hospitalization, no supplements will be prescribed after hospital discharge.

Tested variables will be noted using standard descriptors (arithmetic mean and standard deviation or median). Associations between variables will be assessed using Spearman's rho rank correlation coefficient, the Kruskal-Wallis test for independent samples and a logistic regression model to test statistically significant correlations between PTH and serum calcium values as a primary end point.

ELIGIBILITY:
Inclusion Criteria:

* The patients were eligible if they underwent total thyroidectomy regardless of the surgical indication, if complete serum PTH and calcium data were available through the first five postoperative days and if they signed an informed consent form.

Exclusion Criteria:

* Patients with incomplete data, preoperative pathological calcium or PTH levels, or suffering from conditions affecting calcium metabolism and parathyroid function were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing total thyroidectomy regardless of the surgical indication.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Cut-off PTH post-thyroidectomy value | 5 days
  Statistically significant correlation between postoperative PTH and serum calcium values

SECONDARY OUTCOMES:
Administration of postoperative calcium supplement therapy | 5 days
  Whether or not, and the amount of postoperative calcium supplement therapy needed in case of hypocalcemia

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Rašić, MD, PhD, Study Chair — Department of Otorhinolaryngology and Head and Neck Surgery
Locations (1):
- University Hospital Center Sestre milosrdnice, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No